CLINICAL TRIAL: NCT06598384
Title: Venetoclax Combined With Azacytidine as Maintenance Therapy Post Allogeneic Hematopoietic Stem Cell Transplantation in Myelodysplastic Syndromes and Acute Myeloid Leukemia
Brief Title: VA as Maintenance Therapy Post Allo-HSCT in MDS and AML
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Navy General Hospital, Beijing (Other)
Responsible Party: Principal Investigator, Liren Qian, Vice Director, Navy General Hospital, Beijing
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VAMHCT01
Record Dates: First submitted 2024-09-13; First posted 2024-09-19 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Venetoclax combined with Azacytidine (Experimental): Patients were treated by venetoclax and azacytidine
  Interventions: Drug: Venetoclax combined with Azacytidine

INTERVENTIONS:
Drug: Venetoclax combined with Azacytidine — Patients were treated by venetoclax and azacytidine:
  Venetoclax 100mg po qd d1, 200mg po qd d2, 400mg po qd d3-7; Azacytidine 75 mg/m2 subcutaneous injection qd d1-5.
  Other Names: VA

SUMMARY:
The goal of this phase 2 trial is to test the safety and efficacy of Venetoclax combined with Azacytidine as Maintenance Therapy post Hematopoietic Stem Cell Transplantation in Myelodysplastic Syndromes and Acute Myeloid Leukemia.

DETAILED DESCRIPTION:
The investigators will evaluate the efficacy and safety of venetoclax combined with azacytidine as maintenance therapy post hematopoietic stem cell transplantation in myelodysplastic syndromes and acute myeloid leukemia. overall survival (OS), cumulative 1-year relapse- and progression-free survival (RPFS), time to relapse, relapse rate, incidence of acute and chronic GVHD, time to treatment discontinuation will be counted.

ELIGIBILITY:
Inclusion Criteria:

* The patient should, in the investigator's opinion, be able to meet all clinical trial requirements.
* The patient is willing and able to adhere to the study visit schedule and other protocol requirements.
* Patients aged ≥18 years with a diagnosis of MDS or AML according to World Health Organization criteria (WHO) who had undergone alloSCT with myeloablative or reduced-intensity conditioning regimens were eligible. Related and unrelated donors were permitted.
* Patients should be in morphologic complete remission (CR; ie, ≤5% bone marrow blasts) with absolute neutrophil counts ≥1.0×10^9 /L and platelets ≥ 75×10^ 9 /L before treatment.

Exclusion Criteria:

* Active or uncontrolled infections requiring systemic treatment within 14 days before enrollment.
* Any instability of systemic disease, including but not limited to severe cardiac, liver, kidney, or metabolic disease need therapy.
* Pregnant or lactating women.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2030-09 (Estimated); Study Completion 2030-09 (Estimated)

PRIMARY OUTCOMES:
Relapse Rate | 1 year
  Relapse following CR is defined as reappearance of leukemic blasts in the peripheral blood or the finding of more than 5% blasts in the BM, not attributable to another cause (eg, BM regeneration after consolidation therapy) or extramedullary relapse.

SECONDARY OUTCOMES:
Overall Survival (OS) | through study completion, an average of 2 years
  OS was defined as time from diagnosis to death from any cause or the last follow-up
Progression Free Survival (PFS) | 1 year
  For patients in morphologic remission, documented relapse was considered progression. Relapse following complete remission(CR) is defined as reappearance of leukemic blasts in the peripheral blood or the finding of more than 5% blasts in the BM, not attributable to another cause (eg, BM regeneration after consolidation therapy) or extramedullary relapse.

CONTACTS AND LOCATIONS:
Overall Officials: Liren Qian, Principal Investigator — Navy General Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No